CLINICAL TRIAL: NCT06805370
Title: Randomized Trial of Additional Mailed FIT Kits
Brief Title: Additional Mailed FIT Kits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Mireille Jacobson, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CCHS-QIP-SECOND-FIT-KIT
Record Dates: First submitted 2025-01-15; First posted 2025-02-03 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer Screening
Keywords: fecal immunochemical test (FIT); cancer screening

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Annual FIT Kit Only) (Active Comparator): This arm was sent an annual FIT Kit but was not sent a follow-up FIT Kit in November 2024.
  Interventions: Other: Usual Care
- Mailed Additional FIT Kit (Experimental): This arm was sent a follow-up FIT Kit in November 2024 in addition to the annual FIT Kit mailing.
  Interventions: Behavioral: Mailed Additional FIT Kit

INTERVENTIONS:
Behavioral: Mailed Additional FIT Kit — Mailed additional FIT Kits in November 2024.
  Arms: Mailed Additional FIT Kit
Other: Usual Care — This group was sent an annual FIT Kit per usual care.
  Arms: Usual Care (Annual FIT Kit Only)

SUMMARY:
This study aims to assess whether sending patients in a county health care system additional FIT Kits can increase the FIT Kit return rate enough to warrant the extra cost. To do this, the health system mailed a random subset of patients ages 60 to 75 a FIT Kit in November 2024 in addition to sending patients an annual FIT Kit mailing. This work analyzes the return rate of mailed FIT Kits within 60-days of the November mailing.

DETAILED DESCRIPTION:
This study aims to assess whether sending patients in a county health care system additional FIT Kits can increase the FIT Kit return rate enough to warrant the extra cost. To do this, patients ages 60 to 75 due for colorectal cancer screening, who had not received a FIT Kit in the previous 3 months but had completed one sometime in the past and had an assigned primary care provider, were randomized to be sent a FIT Kit in November of 2024 or to usual care. Usual care includes an annual FIT Kit mailing. We will analyze the successful return rate of mailed FIT Kits within 60-days of the November mailing.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-74
* Due for colorectal cancer screening;
* Not sent a FIT Kit in the past 3-months;
* Previously successfully returned a FIT Kit.

Exclusion Criteria:

* Under age 60 or over age 74;
* Incarcerated;
* Not due for colorectal cancer screening;
* Sent a FIT Kit in the past 3-months.

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
FIT Kit return rate | 60-Days
  Indicator of whether a patient successfully returned a FIT Kit to the health system for processing

CONTACTS AND LOCATIONS:
Locations (1):
- Contra Costa Health, Martinez, California, United States

IPD SHARING:
Plan to Share IPD: No
Researchers can apply for permission to use anonymized data from CCHS.